CLINICAL TRIAL: NCT01721239
Title: Recovery and Aftercare in Post Intensive Care Therapy Patients - The RAPIT Study. The Effectiveness and Experiences of a Follow-up Program for Danish Mechanically Ventilated ICU Patients: A Pragmatic Randomized Controlled Multicentre Trial.
Brief Title: Recovery and Aftercare in Post Intensive Care Therapy Patients - RAPIT Study
Acronym: RAPIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hillerod Hospital, Denmark (Other)
Collaborators: Herlev Hospital (Other); Rigshospitalet, Denmark (Other); Nykøbing Falster County Hospital (Other); Odense University Hospital (Other); Sonderborg Hospital (Other Government); Region of Southern Denmark (Other); Regionshospitalet Horsens (Other); Naestved Hospital (Other)
Responsible Party: Principal Investigator, Janet Froulund Jensen, PHD, MSc Health Science, RN., Hillerod Hospital, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HIH-01863-2012-011
Record Dates: First submitted 2012-10-31; First posted 2012-11-05 (Estimated); Last update posted 2018-04-04 (Actual); Status verified 2018-04

CONDITIONS: Intensive Care (ICU) Patients
Keywords: ICU; Follow-up consultations; Quality of life; Sense Of Coherence; RCT multicenter study

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (No Intervention): No intervention
- Standardized Followup program (Experimental): Standardized written information, patient photos and three follow-up consultations.
  Interventions: Other: Standardized Followup program

INTERVENTIONS:
Other: Standardized Followup program — Standardized written information, patient photos and three followup consultations.
  Arms: Standardized Followup program

SUMMARY:
In 2010 alone were admitted 33,361 patients for treatment in Danish intensive care units. There is evidence to former intensive care patients have a significant symptom burden that affect recovery, function and activity for up to several years after admission to the intensive care unit. For the individual patient involves the low quality of life, delayed recovery, prolonged illness and healing process, and increased mortality. It requires that health professionals should provide support so patients quicker return to their usual life. Follow-up interviews with the staff after hospitalization in ICU have been shown to support the patient and identify individual needs and symptoms that can lead to more realistic expectations and increased well-being after admission in ICU. Follow-up in Denmark is being inconsistent in both the number of hospitals that offer this service, and in the offered type of service. Follow-up interviews with and without diaries suggest to improve physical and mental well-being and health, with limited scientific evidence of the efficacy of these interventions. We will investigate the effect of a standardized follow-up program after admission to the intensive care unit, consisting of written information, patient photos taken during hospitalization and three follow-up calls compared with standard care (discharge without follow-up).

During a clinical study conducted in several intensive care units in Denmark examined whether follow-up calls can improve patients' well-being and health, as well as the meaning of the follow-up program has on the patient's everyday life in the first year after hospitalization in the ICU.

The investigation contribute knowledge to the international research by revealing symptom burden and efficacy of a follow-up program for up to 1 year after admission to the ICU in order to be able to target rehabilitation efforts and improved the quality of life. It will be innovative to use the results from a clinical study as a foundation for a database, and the method can serve as a precedent for evidence-based introduction of guidelines, database registration and create the groundwork for future research in intensive care. This study is expected to be profitable to society by preventing frequent readmissions, reduce medication costs and fewer referrals to specialists and have a positive effect on retention to the labor market. This will provide overall better use of society's expenses.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Non-invasive or invasive ventilation ≥ 48 hours (Non-invasive ventilation (NIV) from current guidelines).
* APACHE II score ≥ 12 ≤ 29
* Unrecognized dementia diagnosis

Exclusion Criteria:

* Delirium at randomization (Positive CAM-ICU score)
* Participation in scientific projects which include patient interviews
* Not Speak and understand Danish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2012-12-01 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Quality of Life | 12 months
  Changes over time in patients in the intervention and control group measured with instruments used and register data, corresponding to quality of life, on the mental component of the instrument, SF-36 Intension-to-treat analysis

SECONDARY OUTCOMES:
Symptom Scores | 12 months
  Changes in score regarding symptoms scores in control and intervention groups.
Baseline data | At randomization
  baseline data concerning patient's demographic and clinical data
Symptom score | 12 months
  Changes over time in patients in the intervention and control group measured with instruments used and register data, corresponding to symptom scores.
Depression | 12 months
  Changes in score regarding depression in control and intervention groups
Sense of Coherence | 12 months
  Changes over time in patients in the intervention and control group measured with instruments used and register data, corresponding to sense of coherence

OTHER OUTCOMES:
Post traumatic stress | 12 months
  Changes in score regarding post traumatic stress in control and intervention groups.
Anxiety | 12months
  Changes in score regarding anxiety in control and intervention groups.
Register data | 12 months
  Changes in score regarding register data concerning:
  1. Mortality
  2. The number of readmissions
  3. Outpatient visits
  4. Referrals to specialists, physical and occupational therapy, including in control and intervention groups
Non-respondent | 12 months
  A non-respondent analysis. The number of participants who dropout of the study will be separated, analyzed in control and intervention groups regarding demographic and clinical data collected during ICU stay. Investigate if there is difference in dropout in the interventiongroup versus the controlgruop.
  Intension-to-treat analysis of participants recieving the first consultation.

CONTACTS AND LOCATIONS:
Overall Officials: Janet F Jensen, PhD-student, Principal Investigator — Hillerod Hospital, department of Anaesthesiology
Locations (1):
- Department of Anaestesiology, Hillerød, Denmark

REFERENCES:
- [Derived] Jensen JF, Egerod I, Bestle MH, Christensen DF, Elklit A, Hansen RL, Knudsen H, Grode LB, Overgaard D. A recovery program to improve quality of life, sense of coherence and psychological health in ICU survivors: a multicenter randomized controlled trial, the RAPIT study. Intensive Care Med. 2016 Nov;42(11):1733-1743. doi: 10.1007/s00134-016-4522-1. Epub 2016 Sep 30. PMID 27695894
- See also: Homepage for project collaborators, this requires departmental access and password — http://posticu.wordpress.com